CLINICAL TRIAL: NCT04588142
Title: Impact of Probiotic Supplementation on Exercise Endurance Among Non-elite Athletes: A Randomized, Placebo-controlled, Double-blind, Clinical Trial
Brief Title: Impact of Probiotic Supplementation on Exercise Endurance Among Non-elite Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: L-020
Record Dates: First submitted 2020-10-01; First posted 2020-10-19 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Exercise Endurance
Keywords: Ergogenic effects; Probiotics; Non-elite athletes
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants are randomized to receive probiotics for 6 weeks
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Participants are randomized to receive placebo for 6 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Non-elite athletes receive probiotic for 6 weeks
  Arms: Experimental group
Dietary Supplement: Placebo — Non-elite athletes receive placebo for 6 weeks
  Arms: Placebo group

SUMMARY:
The aim of this trial is to evaluate the effects of 6-week administration of probiotics on running performance among non-elite athletes. It is hypothesized that participants receiving probiotics may improve their running performance at an endurance test compared to their placebo-receiving counterparts.

DETAILED DESCRIPTION:
Participants recruited from the university community in the Southeast U.S. will participate in a randomized, double-blind, placebo-controlled interventional study for approximately 9 weeks following obtainment of informed consent. Two weeks prior to randomization participants will begin the pre-baseline period and complete daily and weekly questionnaires (physical activity and muscle soreness, bowel movements and gastrointestinal health, flu and cold symptoms). Visit 2 will occur during the pre-baseline period and participants will complete a VO2 max fitness assessment, which will be used during the endurance testing. Participants will also receive the SenseWear Armdand Mini®, a wearable device that will record their physical activity, sleeping patterns and energy expenditure for one week prior to visits 3 and 4.

Participants will be randomized at visit 3. Prior to this visit, participants will consume a standardized breakfast, collect a stool sample and a saliva sample that will be brought to site. During this visit participants will have a body composition and perform the Submaximal Treadmill Test. During the treadmill test, participants will provide finger prick samples for subsequent analysis of blood metabolites (glucose and lactate) and perceived exhaustion subjectively. Lastly, participants will complete several nutrition and motivation-related questionnaires.

One week prior to the final visit (V4), participants will be asked to wear the SenseWear Armband Mini® again for one week, which they will return at the final visit. Participants will eat another standardized breakfast prior to the final visit, visit 4. They will bring a stool and saliva sample to the site. During visit 4, participants will complete the submaximal treadmill test, while providing finger prick samples for analysis of blood and lactate levels. In addition, body composition will be assessed, as well as nutrition and motivation (subjectively). Visit 4 will be followed by a washout week, during which participants will not intake the study supplement but they will complete daily, weekly, and the final questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults between 18-45 years old
2. Regularly participate in running and cross-training, and willing to maintain this level of training throughout the study. Participant must satisfy all three sub-criteria:

   1. 3-5 days per week of running or cross-training AND
   2. 45 minutes - 1.5 hours per activity session AND
   3. Run ≥15 miles per week
3. VO2 max values that in the 60-85th percentile (good-excellent health) range according to ACSM guidelines [1].

Exclusion Criteria:

1. Any physician-diagnosed diseases that would impact exercise performance or participation, including gastrointestinal disease, heart/cardiopulmonary disease, diabetes, thyroid disease, hypogonadism, hepatorenal disease, musculoskeletal disorder, neuromuscular/neurological disease, autoimmune disease, cancer, peptic ulcers or anemia.
2. Professional or elite athletes.
3. Use of any antibiotic drug within 4 weeks of randomization. Volunteer could be eligible to participate after a 2-week washout period.
4. Currently smoking (including vaping)
5. Pregnant, planning to get pregnant, or currently breastfeeding.
6. Lactose intolerance and/or milk, soy or yeast allergy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Time-to exhaustion during submaximal treadmill test | 6 weeks
  Comparison of time-to exhaustion during submaximal treadmill test at the end of intervention from those that received probiotic versus placebo.

SECONDARY OUTCOMES:
Change in perceived exertion | 6 weeks
  Change from baseline in the Borg Rating of Perceived Exertion among probiotics versus placebo (score range = 9, very light effort to 20, extremely strenuous exercise)
Change in blood glucose | 6 weeks
  Change from baseline in capillary blood glucose among probiotics versus placebo
Change in blood lactate | 6 weeks
  Change from baseline in capillary blood lactate among probiotics versus placebo
Difference in salivary stress and immune biomarkers | 6 weeks
  To compare the difference in salivary cortisol, alpha-amylase and sIgA at the end of intervention among probiotics versus placebo
Difference in cold/flu episodes | 6 weeks
  To compare severity, duration and number of cold/flu episodes throughout the intervention among probiotics versus placebo, as assessed by a Visual Analogue Scale
Difference in gastrointestinal function and discomfort | 6 weeks
  To compare GI function during the intervention and change in GI function from baseline among probiotics versus placebo assessed by the Gastrointestinal Symptom Rating Scale (GSRS) and the Digestion-Associated Quality of Life (DQLQ).
Difference in bowel habits | 6 weeks
  To compare bowel habits during the intervention, frequency and consistency, among probiotics versus placebo assessed by the Bristol Stool Form Scale (BSFS)

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, Ph.D., Principal Investigator — University of Florida
Locations (1):
- UF Health Sports Performance Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
After publications of the results, de-identified data will be shared with qualified researchers and scientists upon reasonable request to the sponsor including a detailed proposal of the intended use of the data, as per the Lallemand Health Solutions Inc. Policy on Clinical Trial Transparency and Data Sharing (available upon request).

REFERENCES:
- [Derived] McDermott CE, Vincent HK, Mathews AE, Cautela BG, Sandoval M, Tremblay A, Langkamp-Henken B. Impact of probiotic supplementation on exercise endurance among non-elite athletes: study protocol for a randomized, placebo-controlled, double-blind, clinical trial. Trials. 2022 Jul 27;23(1):603. doi: 10.1186/s13063-022-06552-x. PMID 35897037